CLINICAL TRIAL: NCT07283913
Title: UltraSONIC Vagus Nerve Stimulation: Investigation U-VNS Effects on Physiological, Emotional and Cognitive Biomarkers
Brief Title: Non-invasive Ultrasonic Auricular Vagus Nerve Stimulation
Acronym: SONIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: FMHS 88-0225
Record Dates: First submitted 2025-10-06; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-09

CONDITIONS: Healthy Participants
Keywords: ultrasound vagus nerve stimulation; U-VNS; glucose sensor; health volunteers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active U-VNS (Active Comparator): Participants receive ultrasound vagus nerve stimulation (U-VNS) applied transcutaneously to the cervical vagus nerve using focused ultrasound.
  Interventions: Device: Ultrasound Vagus Nerve Stimulation (U-VNS)
- Sham U-VNS (Sham Comparator): Participants undergo the same procedure with identical setup and audible sound cues, but no ultrasound energy is delivered.
  Interventions: Device: Ultrasound Vagus Nerve Stimulation (U-VNS)

INTERVENTIONS:
Device: Ultrasound Vagus Nerve Stimulation (U-VNS) — 30 minutes of U-VNS delivered to the left auricular branch of the vagus nerve via NeurGear ZenBud vagus nerve stimulator applied to the left ear.

SUMMARY:
The Vagus nerve, one of 12 cranial nerves that connect the brain to the human body, controls specific involuntary functions such as breathing, heart rate, the digestive system and the immune system, and it is crucial to unlocking the relaxation response (parasympathetic nervous system).

Vagus nerve stimulation (VNS) can be invasive or non-invasive, and both methods have been trialled in research studies. Some non-invasive VNS involves the use of a device which is placed on the skin, to send electrical impulses to the Vagus nerve. The device sends electrical impulses to some areas of the brain which changes brain activity and helps in treating certain disorders. Invasive methods utilise a surgically implanted Vagus nerve stimulator on the left Vagus nerve in the neck area.

VNS is used in treatment of epilepsy and studies has shown to have a therapeutic effect on treatment resistant depression. Currently, research indicates that invasive VNS to treat anxiety yield mixed results, whilst other studies suggest that VNS with exposure-based therapies might enhance outcomes for anxiety patients.

Stimulating the Vagus nerve comes with serious technical challenges. Most importantly, electric currents follow the path of least resistance. When running through biological tissues, such as skin, cartilage or bone, it is difficult to aim for the part of the body that needs to be stimulated. This means it isn't always easy to tell whether the Vagus nerve is indeed being stimulated and how much of the current is reaching the Vagus nerve.

This problem can be overcome by ultrasound stimulation. Ultrasound stimulation employs high frequency sound waves to stimulate tissue. These soundwaves travel through the human body much more predictably than electric currents. As such, ultrasound stimulation of the Vagus nerve may be more effective than electrical stimulation. The ZenBud device is designed to apply ultrasound stimulation to part of the auricular branch of the Vagus nerve. Ultrasound stimulation allows for more targeted stimulation, increasing the chance of the stimulation reaching the Vagus nerve. The ZenBud device is safe for use in healthy adults and received CE marking.

Before testing the therapeutic effect of the Zenbud on patients with symptoms it is important to identify physiological, cognition or emotional changes in health volunteers. Identifying these changes could lead to identifying possible future therapeutic uses for ultrasound-VNS (U-VNS).

DETAILED DESCRIPTION:
The vagus nerve is the longest cranial nerve travelling from the medulla to the colon and is involved in the autonomic, cardiovascular, respiratory, gastrointestinal, immune and endocrine systems. The vagus nerves are part of the body's nervous system and control specific bodily functions such as mood, breathing and heart rate, the digestive system and immune system. These responses are involuntary and are not controlled consciously. The vagus nerve is one of twelve cranial nerves that connect the brain to the body. It runs from the brain stem into the gut and is part of the rest and digest system, crucial to unlocking the relaxation response of the parasympathetic nervous system.

Vagus nerve stimulation (VNS) is established as a therapeutic treatment for epilepsy and has promise as a treatment in neuropsychiatric conditions such as drug-resistant depression and headaches. Stimulation of the vagus nerve can be conducted either invasively via a surgical implant or non-invasively (transcutaneous). Transcutaneous VNS can be delivered via the ear, stimulating the auricular branch of the vagus nerve, or at the neck, stimulating the cervical branch. Invasive VNS entails the implantation of a pulse generator device connected to electrodes placed around the cervical vagus nerve; implantation can lead to infection around the wound site, pain, and peri-incisional haematoma.

Traditionally, VNS is electrical, which presents technical limitations since stimulating currents are conducted differently depending on the tissue, and controlling the focus and direction of the current is challenging as it diffuses. In tVNS it is impossible to determine with absolute certainty whether, and to what extent, the administered electric current reaches the vagus nerve.

Ultrasound stimulation of the vagus nerve is an alternative to electrical stimulation through the employment of high-frequency sound waves, which stimulate the central nervous system. The ZenBud device uses ultrasound stimulation on the vagus nerve branch that runs through the ear region. Applying pulses rather than an electric current overcomes technical issues related to electrical conductivity. Ultrasound stimulation enables targeted activation, increasing the likelihood that the stimulation reaches its intended site. ZenBud devices are evidenced as safe to use among healthy adults and have received CE marking following assessments conducted at the University of Nottingham.

Anatomical studies propose that direct stimulation of the vagus nerve fibres in the ear region can produce similar effects to invasive VNS and reduce somatic symptoms of mild to moderate depression and epilepsy, avoiding the need for surgery, which is a common feature of invasive VNS. The presence of tVNS has been associated with improvements in psychological wellbeing. Animal studies suggest that stimulation of the ear area and its vagus nerve fibres produces physiological changes such as decreased heart rate and arterial pressure. Studies have shown that VNS can be effective in treating epilepsy and depression, and there is evidence that it may be useful in pain management and autoimmune or inflammatory disorders; however, a greater understanding of its effects on the body is required.

Research indicates that auricular vagus nerve stimulation can influence EEG and EMG activity in healthy individuals and suggests potential as a non-invasive treatment for various clinical conditions.

The purpose of this study is to investigate the efficacy, safety and usability of the wearable headset and to identify changes in biomarkers due to the use of ultrasound VNS. Identifying physiological, cognitive or emotional changes could help determine potential future therapeutic uses for U-VNS.

For this study, participants will attend multiple visits, with an upper limit of five. Participants will be randomly allocated to receive either U-VNS in the first appointment and sham in the second, or vice versa. Sham will consist of wearing the device without stimulation being delivered.

At the first appointment, safety screening will be confirmed using the U-VNS safety questionnaire, and informed consent will be obtained. Participants will have heart rate and blood pressure recorded. Then, participants will insert a continuous glucose monitor (CGM, Dexcom) and be given a Fitbit smartwatch to wear for monitoring physiological signals, activity and sleep throughout the study.

For the second appointment, participants will be asked to avoid exercise and fast from food for 12 hours prior to arrival. Physiological (heart rate and blood pressure), cognitive and emotional markers will be recorded. A pre-, during- and post stimulation ECG may be performed. EEG data may also be recorded before, during and after stimulation on the same day. Additional physiological markers such as body temperature, skin conductance (via GSR), or ear electrodes located on the cymba conchae through a bipolar electrode may also be recorded.

Participants will complete questionnaires about emotional wellbeing and sleep, such as the STAI and a short Oxford-Liverpool Inventory of Feelings and Experiences (O-Life) and undergo cognitive assessments. These tasks will be completed using PsychoPy or a similar application and will focus on attention, emotion and memory. All tasks involve visual stimuli with responses recorded via keyboard or mouse, and each takes approximately 5-10 minutes to complete. These tasks provide a comprehensive assessment of cognitive and emotional functioning and are tailored to measure domains influenced by VNS.

Following this, participants will receive the intervention using the ZenBud or sham device for up to 30 minutes. After 30 minutes, the device will automatically turn off. Participants will again complete the physiological, cognitive and emotional assessments 10 minutes after stimulation onset and after completion. The participants will also complete the effectiveness of blinding and adverse effects questionnaires.

After a one-week washout period, participants will attend a third appointment. Participants will be asked about any eligibility changes and confirm continued consent. As in the second appointment, participants will fast and refrain from exercise for 12 hours before undergoing the alternate intervention (U-VNS or sham) for 30 minutes. The same assessments and questionnaires will be repeated.

During the second and third visits, participants will use the ZenBud device for up to 30 minutes. If the participants received real U-VNS first, the participants will receive sham second, and vice versa. The device automatically turns off after 30 minutes.

Apart from collecting demographics and medical history during the first visit, the second and third visits will include the same physical, cognitive and emotional assessments before, during and after U-VNS. Participants will wear a Fitbit throughout the study to monitor heart rate and sleep patterns

ELIGIBILITY:
Inclusion Criteria

* Participant is willing and able to give informed consent for participation in the study
* Not currently taking any medications (except the contraceptive pill)
* Aged 18 or over
* Good general health
* Able and willing to remove any piercings in the left ear
* Able to abstain from exercise and fast from food for 12 hours before the second and third visit

Exclusion Criteria

* Current or past diagnosis of a major neurological, neurosurgical, or psychiatric disorder (including self-reported depression)
* Inability to complete informed consent process
* Personal history of cardiac arrhythmia
* Diabetes
* High blood pressure (>140 mmHg systolic and/or >90 mmHg diastolic)
* Other significant medical condition (including cardiological disorders; specific details to be reviewed by the CI prior to inclusion)
* Use of medication or recreational drugs that affect the nervous system in the past 3 months
* Medication intake (such as beta-blockers, glucocorticoids, antidepressants, anti-inflammatory drugs) in the last 7 days - contraceptive medication in women is allowed
* Currently pregnant or breastfeeding
* Allergy to aquasonic gel or any of its components (propylene glycol, glycerin, isothiazolinones)
* Participation in a research study in the last 3 months involving invasive procedures or an inconvenience allowance (required for all UoN FMHS UREC-approved studies)
* BMI < 18 kg/m² or > 30 kg/m²
* Excessive consumption of alcohol (>2 alcoholic beverages/day) or tobacco (>5 cigarettes/day)
* Previous experience with stress tests
* Known infection in the last 8 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Continuous Glucose Monitoring (CGM)-derived glycaemic variability | Baseline to 20-25 days. Measurements taken every 5 minutes continuously through a GCM device. Measurements taken in mg/dL
Glucose Level measured in mg/dL extracted derived from Continuous Glucose Monitoring (CGM) | Baseline to 20-25 days with Baseline to 20-25 days. Measurements taken every 5 minutes continuously through a GCM device. Measurements taken in mg/dLin between
EEG Power in Alpha Band (8-12Hz) | Baseline to 20-25 days, measured before, during, and after stimulation
EEG Power in Theta Band (4-7Hz) | Baseline to 20-25 days, measured before, during, and after stimulation
EEG Power in Beta Band (13-30Hz) | Baseline to 20-25 days, measured before, during, and after stimulation
EEG Power in Gamma Band (31-45Hz) | Baseline to 20-25 days, measured before, during, and after stimulation
EEG-derived Event-Related Potential (ERP) amplitude | Baseline to 20-25 days, measured before, during, and after stimulation
EEG-derived Time-locked spectral power changes | Baseline to 20-25 days, measured before, during, and after stimulation
ECG-derived Heart Rate (HR) | Baseline to 20-25 days, measured before, during, and after stimulation
ECG-derived QT interval | Baseline to 20-25 days, measured before, during, and after stimulation
ECG-RR Interval (inter-beat Interval) | Baseline to 20-25 days, measured before, during, and after stimulation
ECG-derived Heart Rate Variability (HRV) | Baseline to 20-25 days, measured before, during, and after stimulation
ECG-derived PR Interval | Baseline to 20-25 days, measured before, during, and after stimulation

SECONDARY OUTCOMES:
Fitbit smartwatch-derived Heart Rate (HR) during sleep | Baseline to 20-25 days. Measurements taken continuously through a Fitbit device with PPG
Fitbit smartwatch-derived Daily Heart Rate Variability (HRV) | Baseline to 20-25 days. Measurements taken continuously through a Fitbit device with PPG
Fitbit smartwatch-derived resting Heart Rate (HR) | Baseline to 20-25 days. Measurements taken continuously through a Fitbit device with PPG
Fitbit smartwatch-derived daily step count | Baseline to 20-25 days. Measurements taken continuously through a Fitbit device
Fitbit smartwatch-derived daily ratio of Sedentary (no activity) vs active time | Baseline to 20-25 days. Measurements taken continuously through a Fitbit device
Fitbit smartwatch-derived Total sleep duration (hours per day) | Baseline to 20-25 days. Measurements taken continuously through a Fitbit device
Fitbit smartwatch-derived daily percentage of sleep stages (including light, deep and REM sleep) | Baseline to 20-25 days. Measurements taken continuously through a Fitbit device.
Fitbit smartwatch-derived daily sleep efficiency measured as daily ratio of total sleep time to time in bed | Baseline to 20-25 days. Measurements taken continuously through a Fitbit device
Continuous Skin conductance (electrodermal activity) levels measured via GSR sensors (kOhms) | Baseline to 20-25 days, measured before, during, and after stimulation
Continuous Body temperature measured using a thermistor (°C) | Baseline to 20-25 days, measured before, during, and after stimulation
Respiration Rate measured as percentage of chest expansion (%) through a wearable chest sensor | Baseline to 20-25 days, measured before, during, and after stimulation
Vagus Nerve electrical activity (µV) variability recorded through a bipolar electrode placed on the cymba conchae of the right ear. | Baseline to 20-25 days, measured before, during, and after stimulation
Event-related Vagus Nerve amplitude changes recorded through a bipolar electrode placed on the cymba conchae of the right ear | Baseline to 20-25 days, measured before, during, and after stimulation
Total score on the Oxford-Liverpool Inventory of Feelings and Experiences questionnaire. Higher scores indicate higher levels of schizotypal traits. | Baseline, questionnaire done once before the first visit
Total score on the Autism-Spectrum Quotient (AQ) questionnaire. Higher scores indicate greater or higher presence of autistic traits. | Baseline, questionnaire done once before the first visit
Total score on the Multidimensional Assessment of Interoceptive Awareness (MAIA) questionnaire. Higher scores indicate greater interoceptive awareness. | Baseline, questionnaire done once before the first visit
Total score on the State-Trait Anxiety Inventory - Trait subscale (long form). Higher scores indicate greater trait anxiety. | Baseline, questionnaire done once before the first visit
Total score on the State-Trait Anxiety Inventory - Trait subscale (short form). Higher scores indicate greater state anxiety. | Baseline to 20-25 days, questionnaire done before the first visit, one hour before stimulation and one hour after stimulation
Total score on the Beck Depression Inventory (range 0-63). Higher scores indicate more severe depressive symptoms | 24 hours after stimulation
Total score on the Beck Anxiety Inventory (BAI) (range 0-63). Higher scores indicate more severe anxiety symptoms. | 24 hours after stimulation
Structured questionnaire assessing adverse effects of ultrasonic Vagus nerve stimulation (VNS). | 24 hours after stimulation
Average Reaction time (ms) measured from a Stroop Cognitive task | Baseline to 20-25 days, measured immediately before, during, and immediately after stimulation
Average Reaction time (ms) measured from a Semantic Memory Cognitive task | Baseline to 20-25 days, measured immediately before, during, and immediately after stimulation
Average Reaction time (ms) measured from an Emotional Bias Cognitive task. | Baseline to 20-25 days, measured immediately before, during, and immediately after stimulation
Average Reaction time (ms) measured from a symbol-to-symbol matching Cognitive task. | Baseline to 20-25 days, measured immediately before, during, and immediately after stimulation
Average Reaction time (ms) measured from an Object-in-place Working memory Cognitive task | Baseline to 20-25 days, measured immediately before, during, and immediately after stimulation
Overall task accuracy (%) measured from a Stroop Cognitive task. | Baseline to 20-25 days, measured immediately before, during, and immediately after stimulation
Overall task accuracy (%) measured from a Semantic Memory Cognitive task | Baseline to 20-25 days, measured immediately before, during, and immediately after stimulation
Overall task accuracy (%) measured from an Emotional Bias Cognitive task. | Baseline to 20-25 days, measured immediately before, during, and immediately after stimulation
Overall task accuracy (%) measured from a symbol-to-symbol matching Cognitive task | Baseline to 20-25 days, measured immediately before, during, and immediately after stimulation
Overall task accuracy (%) measured from an Object-in-place Working memory Cognitive task. | Baseline to 20-25 days, measured immediately before, during, and immediately after stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Kaiser, Professor, Principal Investigator — University of Nottingham; Amparo G Gonzalez, PhD, Principal Investigator — University of Cambridge
Locations (2):
- United Kingdom (2):
  - Neuromodulation Lab, Medical School, Queen's Medical Centre, Nottingham, Nottinghamshire
  - University of Nottingham, Nottingham

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Colzato L, Beste C. A literature review on the neurophysiological underpinnings and cognitive effects of transcutaneous vagus nerve stimulation: challenges and future directions. J Neurophysiol. 2020 May 1;123(5):1739-1755. doi: 10.1152/jn.00057.2020. Epub 2020 Mar 25. PMID 32208895
- [Background] Bartolomei F, Bonini F, Vidal E, Trebuchon A, Lagarde S, Lambert I, McGonigal A, Scavarda D, Carron R, Benar CG. How does vagal nerve stimulation (VNS) change EEG brain functional connectivity? Epilepsy Res. 2016 Oct;126:141-6. doi: 10.1016/j.eplepsyres.2016.06.008. Epub 2016 Jul 29. PMID 27497814
- [Background] Johnson RL, Wilson CG. A review of vagus nerve stimulation as a therapeutic intervention. J Inflamm Res. 2018 May 16;11:203-213. doi: 10.2147/JIR.S163248. eCollection 2018. PMID 29844694
- [Background] Liu RP, Fang JL, Rong PJ, Zhao Y, Meng H, Ben H, Li L, Huang ZX, Li X, Ma YG, Zhu B. Effects of electroacupuncture at auricular concha region on the depressive status of unpredictable chronic mild stress rat models. Evid Based Complement Alternat Med. 2013;2013:789674. doi: 10.1155/2013/789674. Epub 2013 Jan 29. PMID 23431349
- [Background] Henry TR. Therapeutic mechanisms of vagus nerve stimulation. Neurology. 2002 Sep 24;59(6 Suppl 4):S3-14. doi: 10.1212/wnl.59.6_suppl_4.s3. PMID 12270962
- [Background] Butt MF, Albusoda A, Farmer AD, Aziz Q. The anatomical basis for transcutaneous auricular vagus nerve stimulation. J Anat. 2020 Apr;236(4):588-611. doi: 10.1111/joa.13122. Epub 2019 Nov 19. PMID 31742681
- [Background] Toffa DH, Touma L, El Meskine T, Bouthillier A, Nguyen DK. Learnings from 30 years of reported efficacy and safety of vagus nerve stimulation (VNS) for epilepsy treatment: A critical review. Seizure. 2020 Dec;83:104-123. doi: 10.1016/j.seizure.2020.09.027. Epub 2020 Oct 10. PMID 33120323
- [Background] Breit S, Kupferberg A, Rogler G, Hasler G. Vagus Nerve as Modulator of the Brain-Gut Axis in Psychiatric and Inflammatory Disorders. Front Psychiatry. 2018 Mar 13;9:44. doi: 10.3389/fpsyt.2018.00044. eCollection 2018. PMID 29593576
- [Background] Yuan H, Silberstein SD. Vagus Nerve and Vagus Nerve Stimulation, a Comprehensive Review: Part I. Headache. 2016 Jan;56(1):71-8. doi: 10.1111/head.12647. Epub 2015 Sep 14. PMID 26364692
- [Background] Kohler I, Hacker J, Martin E. Reduction of Anxiety-Related Symptoms Using Low-Intensity Ultrasound Neuromodulation on the Auricular Branch of the Vagus Nerve: Preliminary Study. JMIR Neurotechnol. 2025 May 1;4:e69770. doi: 10.2196/69770. eCollection 2025. PMID 41341418